CLINICAL TRIAL: NCT01737216
Title: Pilot Study of Zoledronic Acid in Combination With First-line Chemotherapy in Aged Patients With Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hebei Tumor Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HBTH201; Hebei Tumor Hospital (Registry Identifier: Hebei Tumor Hospital)
Record Dates: First submitted 2012-11-27; First posted 2012-11-29 (Estimated); Last update posted 2012-12-31 (Estimated); Status verified 2012-11

CONDITIONS: Lung Cancer
Keywords: Aged; patients
MeSH Terms: conditions — Lung Neoplasms | interventions — Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Zoledronic acid plus First-line chemotherapy (Experimental)
  Interventions: Drug: Zoledronic acid plus EP/TP
- First-line chemotherapy (Active Comparator)
  Interventions: Drug: EP/TP

INTERVENTIONS:
Drug: Zoledronic acid plus EP/TP — Drug:EP/TP+Zoledronic acid EP(VP-16 100mg/m2 d1-3;DDP 60-75mg/m2 d1) every 4 weeks, for 4-6 cycles TP(PTX 135-175mg/m2 d1;DDP 60-75mg/m2 d1) every 3 weeks, for 4-6 cycles Zoledronic acid 4mg d1 every 3 months until bone metastasis, 4mg d1 every 1 month until progression
  Arms: Zoledronic acid plus First-line chemotherapy
Drug: EP/TP — Drug:EP/TP EP(VP-16 100mg/m2 d1-3;DDP 60-75mg/m2 d1) every 4 weeks, for 4-6 cycles TP(PTX 135-175mg/m2 d1;DDP 60-75mg/m2 d1) every 3 weeks, for 4-6 cycles
  Other Names: First-line chemotherapy
  Arms: First-line chemotherapy

SUMMARY:
Pilot study of Zoledronic acid in combination with first-line chemotherapy in aged patients with lung cancer. The purpose is to assess the effects of Zoledronic acid in combination with first-line chemotherapy in aged patients with lung cancer on bone mineral density gain in the lumbar spine and total hip.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Age ≥70 years
* Performance Status- Eastern Cooperative Oncology Group (ECOG) 0-1
* Histologically or cytologically confirmed lung cancer
* Did not receive bisphosphonate treatment

Exclusion Criteria:

* Appear relapse and metastasis
* receive other bisphosphonate treatment
* Active or uncontrolled infection
* Pregnant or lactating women

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-11; Primary Completion 2016-01 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival(PFS) | 1 year

SECONDARY OUTCOMES:
Overall survival(OS) | 3 years
Bone mineral density(BMD) | 1 year
Quality of life(QOL) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Wei Liu, Principal Investigator — Hebei Tumor Hospital
Locations (1):
- Hebei Tumor Hospital, Shijiazhuang, Hebei, China